CLINICAL TRIAL: NCT06631209
Title: Effectiveness of Transcranial Magnetic Stimulation of the Default Mode Network to Improve Sleep - Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00005073
Record Dates: First submitted 2024-09-20; First posted 2024-10-08 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Insomnia
Keywords: Sleep Quality; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Transcranial Magnetic Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: There will be 4 parallel groups of 30 participants, each receiving either one of the 3 possible stimulation sites or receiving placebo "Sham". The total number of subjects to be recruited locally to complete all study activities will be n=120. Due to prior experience with similar multi-day studies, it is expected that ~20% dropout before completion. Therefore, assuming this dropout rate (i.e., 24 consented participants), the plan is to enroll a total of 144 participants to achieve the final sample of 120 unable datasets.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Active Stimulation - Posterior Cingulate Cortex (Active Comparator): Active Stimulation targeted at the Posterior Cingulate Cortex
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Active Stimulation - Inferior Parietal Lobule (Active Comparator): Active Stimulation targeted at the Inferior Parietal Lobule
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Active Stimulation - Dorsomedial Prefrontal Cortex (Active Comparator): Active Stimulation targeted at the Dorsomedial Prefrontal Cortex
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Sham Stimulation (Sham Comparator): The TMS device will be placed to the head but no energy will be emitted.
  Interventions: Other: Sham

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Specifically, Continual Theta Burst Stimulation
  Arms: Active Stimulation - Dorsomedial Prefrontal Cortex; Active Stimulation - Inferior Parietal Lobule; Active Stimulation - Posterior Cingulate Cortex
Other: Sham — Sham TMS
  Arms: Sham Stimulation

SUMMARY:
The investigators propose to expand our previous work to test whether 10 repeated administrations of the cTBS procedure over a two-week period can lead to longer-term improvements in sleep, perhaps up to 3-months. For this 3-year study, 120 people with insomnia will be recruited to participate. There will be an initial screening, with the first consent form being for the screening questions, a psychological interview, and a one night at home sleep monitoring session with our equipment. If participants pass this first phase, they will reconsent for the main portion of the study. They will then undergo a physical examination, then a week-long at-home monitoring phase where they will wear a wristwatch sleep monitor as well as wear a portable brain wave monitor to bed each night to record sleep. Participants will continue to use this equipment throughout the treatment phase and for one week post treatment. After the first monitoring phase, each participant will be randomly assigned to one of four different conditions (i.e., 30 assigned to each group). Three of the conditions will involve cTBS focused on different brain locations (i.e., stimulation to the middle front, middle back, or side of the skull), while the fourth condition will provide inactive sham stimulation as a control. All participants will complete 10 treatment visits to the lab over two-to-three weeks, during which they will get a brief cTBS or sham stimulation each time. In addition, all participants will complete a brain scanning and cognitive testing session at the beginning and end of the two-to-three week treatment period. Participants will also complete 1-month and 3-month online follow-up assessments to examine long-term effects.

DETAILED DESCRIPTION:
Phase 0: Screening and Rule-Outs:

During the REDCap Screening, participants will first read this informed consent form and sign it electronically on REDCap to proceed. To begin the screening questions, they must pass a 10-question comprehension check with questions regarding this document to ensure you understand the study. They will then answer a series of questionnaires related to demographics and health background. The REDCap screener will automatically end the survey if they indicate any exclusion. If you are included in the study, at the end of the screening questions it will indicate so and that we will be in contact with you shortly. They will then undergo a virtual psychological interview to determine if they indeed have Insomnia to qualify for the study. Then, they will be mailed WatchPAT monitoring equipment for them to utilize for one night of sleep monitoring at home. This device will measure their level of Obstructive Sleep Apnea, excluding them if they score >15 AHI. We will review all of this data, and if they are eligible, participants will move on to Phase 1 of the study and undergo a second consent form.

Phase 1 In-Person Screening/Enrollment, Pre-Intervention:

Individuals who are eligible for this study after the three screening points will come into the lab to undergo an informational briefing and physical screening appointment. At this appointment, potential participants will complete the main consent for the rest of the study and get to ask any additional questions they have in person. Then, they will undergo a physical examination with a physician to determine eligibility. During the physical examination, there will be a collection of vital signs, EKG, and urine samples to screen for pregnancy and drugs (Ketamine, cocaine, MDMA, phenylcycline (PCP), and amphetamines). We will not be excluding for marijuana. In addition, individuals will complete evaluations to assess intelligence and cognition. If an individual is physically eligible and wishes to move forward, they will then be sent home and asked to complete 7 days of at-home sleep monitoring. This will include wearing an actigraph and a MUSE headband every night, while completing daily sleep diaries and short surveys every morning.

Phase-2 Baseline/Randomization/Active Intervention:

At the baseline visit participants will be asked to complete several cognitive and emotional assessments, have a pre-TMS neuroimaging scan and Electrocardiogram session, and undergo their first TMS administration. The first TMS administration will follow participant randomization into one of the four study conditions.

Following the baseline visit, during treatment participants will be asked to continue using the MUSE headband and actigraph every night and complete daily sleep diaries every morning. Participants will also be asked to return to the lab for 10 total TMS sessions in 2-3 weeks, all lasting around an hour in the evening. Participants will be administered a PVT task before and after each treatment session.

The kind of TMS we are administering is called Theta Burst Stimulation (TBS). A MagVenture MagPro X100 stimulator (MagVenture Inc. Denmark) connected with a figure-of-eight magnetic coil with active cooling will be used for the TBS protocol. Each individual is expected to have a different sensitivity to the magnetic fields generated by the cTBS, and the stimulation intensity will need to be adjusted based on each individual's resting motor threshold (RMT). Once we determine the RMT, we will set the machine to run at 70% of this level. The stimulation will last 40 seconds.

The ten TMS sessions will last for one hour between 6-9pm on weekdays. Ideally, there would be a session every weekday straight for two full weeks. We understand that this may be difficult for some people. If you need to miss a day or two, that is okay. However, 10 sessions are required. The maximum administration window is 3 weeks. The maximum number of days you can go between TMS sessions is 4 days. Please refrain from engaging in exercise in the time between your evening TMS session and when you go to bed.

Phase 3- Post-Intervention:

After participants complete the two-to-three-weeks of active intervention they will be asked to return to the lab to complete a post-intervention visit. This will involve the same testing as the pre-intervention (baseline) visit (MRI, surveys, and ECG). After this visit, participants will be sent home to continue recording sleep/activity for 7 more nights with the MUSE headband and actigraph, as well as continue recording sleep diaries and short surveys. This is the same as the at-home visit pre-intervention. After post-monitoring, participants will return to the lab for their final close-out visit. During this visit participants will return all study equipment and that will be the last of the in-person visits.

Phase 4- Follow-Up:

Participants who agree during the consent process will be contacted 1-month and 3-months after study completion to complete a series of brief assessments on REDCap, as well as another Psychological Interview at the 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and non-pregnant women 18-60 (inclusive) years of age free from contraindicated diseases, medications, devices, and conditions.
* Must score in the moderate or higher range on the Insomnia Severity Index (ISI ≥ 15)
* Must meet the criteria for DSM-5 insomnia disorder as determined by a clinical interview with a board-certified sleep medicine physician.
* Sex ratio will be set to ~50% males; ~50% females
* Ethnicity ratio will be set to ~29.5% who identify as a minority; ~70.5% who identify as white

Exclusion Criteria:

* Presence of any metal implant or medical device that may pose a safety risk for MRI or TMS (permanent hearing aids, cochlear implants, medication infusion devices, brain stimulation devices, permanent retainer, etc.)
* Self-reported past or present medical diagnosis of sleep or breathing-related disorders such as sleep apnea other than insomnia (potential confounder);
* Confounder of Obstructive Sleep Apnea as measured by WatchPAT device at home
* Travel outside the time zone within the one week prior to the physical visit and at any point while active in the study (known to affect sleep);
* Regular shiftwork within 6-months prior to enrollment in the study (known to affect sleep);
* Self-reported past or present history of any seizures or seizure disorders or other contraindication to neurostimulation, for self or any first-degree relatives (safety concern);
* Self-reported current use of certain prescription medications that can either influence seizure threshold, or neuroimaging findings (safety concern and potential confounder);
* Self-reported caffeine use in excess of 300 mg (e.g., approximately 8 caffeinated sodas or approximately 3-4 12-oz cups of coffee) per day on average (known to affect sleep; potential confounder);
* Self-reported or suspected substance abuse or dependence (safety concern; potential confounder);
* (Females only) Positive urine pregnancy result (Urine HCG Test results) (safety concern);
* Inability to read and sign the consent form (regulatory/ethical issue)
* Self-reported history of repeated, recent, or severe fainting spell or syncope
* Prior spinal cord surgeries or any spinal/ventricular derivations
* Self-reported negative experience due to neurostimulation before
* Deviation from self-reported normal bedtime sleep schedules (bedtime between 9:00 pm and 1:00 am

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Sleep stage changes as determined by Polysomnography | 1 month
  PSG will be taken nightly during at home monitoring and treatment
Change in scores on the Pre-Sleep Arousal Scale (PSAS) | 4 months
  Scale will be taken daily for main 4 weeks of study and taken again at 1 month and 3 month followup. Total score ranging from 16-80. Two subscores (somatic and cognitive arousal) ranging from 8-40. Higher scores indicating greater arousal
Change in Insomnia Severity Index (ISI) score | 4 months
  Scale will be taken before and after treatment and at followups at 1 month and 3 months. Score ranging from 0-28 with higher scores indicating greater levels of insomnia.
Sleep duration change as determined by Polysomnography | 1 month
  PSG will be taken nightly during at home monitoring and treatment
Sleep efficiency change as determined by Polysomnography | 1 month
  PSG will be taken nightly during at home monitoring and treatment
Sleep latency change as determined by Polysomnography | 1 month
  PSG will be taken nightly during at home monitoring and treatment
Wakefulness after sleep onset (WASO) change as determined by Polysomnography | 1 month
  PSG will be taken nightly during at home monitoring and treatment
Change in DMN within-network connectivity during resting state | 3 weeks
  fMRI data will be collected during resting state in the scanner for pre and post

SECONDARY OUTCOMES:
Change in DMN activity during a cognitively demanding task | 1 week
  fMRI data will be collected during a task in the scanner for pre and post
Change in GABA levels in the posterior cingulate cortex | 3 weeks
  Spectroscopy data will be collected during resting state in the scanner for pre and post
Change in glutamate/glutamine (glx) levels in the posterior cingulate cortex | 3 weeks
  Spectroscopy data will be collected during resting state in the scanner for pre and post
Correlation between changes in GABA/glx levels and changes in resting state functional connectivity within the DMN | 3 weeks
  Spectroscopy and fMRI data will be collected during resting state in the scanner for pre and post
Correlation between changes in GABA/glx levels and changes in functional deactivation of the DMN during a cognitive challenge task | 3 weeks
  Spectroscopy and fMRI data will be collected in the scanner for pre and post
Change in lactate levels in the posterior cingulate cortex | 3 weeks
  Spectroscopy data will be collected during resting state in the scanner for pre and post
Change in dynamic diffusion along the perivascular space | 3 weeks
  Dynamic diffusion data will be collected during resting state in the scanner for pre and post
Change in scores on the Penn State Worry Questionnaire (PSWQ). | 4 months
  Scale will be taken at pre and post treatment, and taken again at 1 month and 3 month followup. Score ranging from 16-80, with higher scores indicating higher levels of worry
Change in scores on the Epsworth Sleepiness Scale (ESS) | 4 months
  Scale will be taken before and after treatment and at 1 month and 3 months follow-ups. Score ranging from 0-24 with higher scores indicating greater sleepiness.
Change in scores on the Functional Outcomes of Sleep Questionnaire (FOSQ) | 4 months
  Scale will be taken before and after treatment and at followups at 1 month and 3 months. Score ranging from 5-20 with lower scores indicating greater life impairment due to sleep.
Change in spectral density measure of the EEG beta1 and beta2 frequency bands with a focus on the frontal electrodes (Fp1, F7, F8) | 1 month
  EEG will be collected every night during at-home monitoring and treatment
Change in sleep duration determined by actigraphy | 1 month
  Actigraphy will be collected nightly during sleep period
Change in sleep efficiency determined by actigraphy | 1 month
  Actigraphy will be collected nightly during treatment and at-home monitoring periods
Change in sleep latency determined by actigraphy | 1 month
  Actigraphy will be collected nightly during treatment and at-home monitoring periods
Change in wakefulness after sleep onset (WASO) as determined by actigraphy | 1 month
  Actigraphy will be collected nightly during treatment and at-home monitoring periods
Change in in Psychomotor Vigilance Task (PVT) performance | 1 month
  PVT will be administered during pre and post MRI and before and after every treatment session.
Change in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 1 month
  RBANS will be administered during pre and post MRI days. The scale score ranges from 40-160, with 100 being the average. Higher scores indicate greater cognitive ability
Changes in sleep as determined by self-report sleep diaries | 1 month
  Sleep diaries will be filled out daily during at-home monitoring and treatment periods. Questions about nightmares, sleep quality, naps, and wake-ups are recorded.
Change in Spielberger State-Trait Anxiety Inventory (STAI) | 4 months
  Taken at pre and post MRI days and at both followups. State and trait scores result, ranging from 20-80 each. Higher scores indicate greater anxiety
Change in Epworth Sleepiness Scale | 4 months
  Taken at both MRI days and at both followups. Total score ranging from 0-25 with higher scores indicating greater sleepiness.
Change in Patient Health Questionnaire - 9 (PHQ-9) | 4 months
  Taken at screener, at pre and post MRI days, and at both followups. Scores ranging from 0-27 with higher scores indicating greater depression
Change in Pittsburgh Sleep Quality Index | 4 months
  Taken at both MRI days and at both followups. Global score ranging from 0-78 and 7 component scores (sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction). Higher scores indicating greater sleep disturbances.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Related Impairment Scale | 4 months
  Taken at both MRI days and at both followups. Score ranging from 8-40 with higher scores indicating more impaired sleep
Change in Patient-Reported Outcomes Measurement Information System - Sleep Disturbance | 4 months
  Taken at both MRI days and at both followups. Score ranging from 8-40 with higher scores indicating more disturbed sleep
Change in Morningness-Eveningness Questionnaire Type | 4 months
  Taken at both MRI days and at both followups. This scale classifies someone as definitely morning type, moderately morning type, neither type, moderately evening type, or definitely evening type.
Change in Glasgow Content of Thoughts Inventory (GCTI) Scale Score | 4 months
  Taken at both MRI days and at both follow-ups. Score ranging from 25-100, with higher scores indicating more intrusive thoughts before sleep.
Change in PTSD Checklist (PCL-5) Score | 4 months
  Taken at both MRI visits and at both follow-ups. Score ranging from 0-80, with higher scores indicating more severe reactions to PTSD
Change in Positive and Negative Affect Schedule (PANAS) Scores | 4 months
  Taken at both MRI visits and followups. A score for positive and a score for negative affect, ranging from 10-50 each. Higher scores in either category indicate a greater amount of that kind of affect.
Change in Nightmare Disorder Index Scores | 4 months
  Taken at both MRI days and at both follow-ups. Score ranging from 0-20 with greater scores indicating more severe nightmares.
Change in Multidimensional Fatigue Inventory Scores | 4 months
  Taken at both MRI days and at both follow-ups. 5 dimensions of fatigue scores ranging from 4-20, one total score ranging from 20-100. Higher scores indicate greater fatigue
Change in Mindful Attention Awareness Scale (MAAS) Score | 4 months
  Taken at both MRI visits and at both follow-ups. Mean score of all items ranging from 1-6, with higher scores indicating greater mindfulness.
Change in Heart Rate Variability (HRV) | 4 weeks
  EKG will be taken at the physical and at both MRI visits. We will determine HRV based off of this data.

CONTACTS AND LOCATIONS:
Locations (1):
- SCAN Lab, Tucson, Arizona, United States